CLINICAL TRIAL: NCT07314905
Title: Adaptive Platform Trial of Treatments for Respiratory Infections in Community Settings
Brief Title: Adaptive Platform Trial of Treatments for Respiratory Infections in Community Settings (TreatResp)
Acronym: TreatResp
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Unity Health Toronto (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Health Canada (Other Government)
Responsible Party: Principal Investigator, Andrew Pinto, Principal Investigator, Unity Health Toronto
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CTO 5178
Record Dates: First submitted 2025-10-01; First posted 2026-01-02 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Influenza A; Influenza B; SAR-CoV-2; Acute Respiratory Infections (ARIs)
Keywords: COVID-19; SARS-CoV-2; Influenza A; Influenza B; Influenza; Respiratory pathogens; Respiratory infections; Adaptative Platform Trials (APT); acute respiratory infections (ARIs)
MeSH Terms: conditions — COVID-19; Influenza, Human; Respiratory Tract Infections | interventions — baloxavir

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Research study staff (Research Assistants, PI, Statistician, QI, Co-PI, Manager and Coordinators)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acute Influenza A/B - Matched placebo for Baloxavir (Placebo Comparator): Usual Care (i.e., supportive care and symptom relief). Matching control placebo for Baloxavir - a single matching dose.
  Interventions: Drug: Placebo Control
- Acute Influenza A/B - Baloxavir (Experimental): The adaptative platform trial will assess therapeutics for influenza A/B in out-patient setting. Interventions include: Baloxavir. Baloxavir dose: if weight <80 kg: one 40 mg dose for 1 day; if weight ≥80kg, one 80 mg dose for one day.
  Interventions: Drug: Baloxavir

INTERVENTIONS:
Drug: Baloxavir — This is a sub-protocol within the TreatResp adaptive platform trial to compare the clinical and cost-effectiveness of Baloxavir, a single 40mg or 80 mg tablet based on patient weight, to a matching placebo among non-hospitalized patients with mild to moderate influenza A/B. This sub-protocol is part of the influenza domain within TreatResp.
  Arms: Acute Influenza A/B - Baloxavir
Drug: Placebo Control — Matching placebo for Baloxavir
  Arms: Acute Influenza A/B - Matched placebo for Baloxavir

SUMMARY:
TreatResp is a double-blind, individually randomized, multi-centre adaptive platform trial. TreatResp aims to establish an adaptive platform trial aimed at evaluating the clinical- and cost-effectiveness, practical challenges, and outcomes of therapeutics for respiratory pathogens in non-hospitalized patients. Participants will be randomized to receive usual care (i.e., supportive care and symptom relief) or a study therapeutic, which will be determined by the TreatResp Therapeutics Committee. The primary outcomes being evaluated is time to recovery.

DETAILED DESCRIPTION:
Effective and affordable therapeutics for respiratory pathogens that can be used easily in community settings are needed to accelerate recovery, prevent hospitalizations and deaths. The Adaptive Platform Trial of Treatments for Respiratory Infections in Community Settings (TreatResp) will evaluate the clinical effectiveness and cost-effectiveness of therapeutics for respiratory pathogens in non-hospitalized patients. Adaptive platform trials (APTs) are designed to compare multiple therapies in an efficient manner and allow us to respond to the dynamic nature of pandemics. Therapeutics to be evaluated will be identified through a transparent TreatResp Therapeutics Committee. The primary outcome is time to recovery (defined as the first instance that a participant report feeling fully recovered), and key secondary outcomes include all-cause emergency department (ED) visit and/or hospitalization and/or death at 28 days, time to sustained resolution, time to progression of signs or symptoms, symptom severity, quality of life, and cost-effectiveness of each therapeutic. TreatResp leverages our CBRF funded Pandemic Preparedness Engaging Primary Care and Emergency Departments (PREPARED) initiative to recruit participants to the study.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* A positive test (PCR or RAT) for one of the pathogens included in the trial's domains (influenza A/B, or other future specified respiratory pathogens),
* Enrolled within 5 days of symptoms onset. However, this window may vary depending on the domain or specific interventions within each domain (for example 72 hours for Baloxavir).
* At least two symptoms commonly associated with respiratory infections, including:

  * rhinitis
  * cough
  * wheezing
  * sore throat
  * nasal congestion
  * shortness of breath
  * fatigue
  * rapid breathing
  * excessive mucus production
  * loss of smell or taste
  * hemoptysis
  * trouble sleeping or insomnia due to breathing difficulties
  * fever (defined for purposes of this study as >37.5°C/ 41).

Exclusion Criteria:

* Admitted to hospital or in an ED for more than 24 hours
* Previously randomized to TreatResp within the past 12 months
* Currently participating in a clinical trial of a therapeutic agent for acute respiratory pathogen infection that is not/suspected not compatible with the study therapeutics
* Already taking a study therapeutic or contraindication to a study therapeutic
* Inability for participant or caregiver to provide informed consent.

Additional eligibility criteria will be applied based on the intervention assigned. For instance, if a participant is randomized to an antiviral treatment, they must not have contraindications specific to that antiviral. This ensures that each treatment is evaluated in a population for whom it is most appropriate and safe.

Baloxavir exclusion:

* Has a known or suspected pregnancy
* Is breastfeeding
* Is of childbearing potential and is not willing to use a highly effective contraceptive
* Has advanced chronic kidney disease (CKD stage 3: eGFR ≥30 to <60 mL/min, and severe renal impairment (eGFR <30 ml/min, CKD stage 4-5)
* Has severe hepatic impairment, or requires a live viral vaccine within the next seven days
* Has a significant impaired immunity (e.g., due to long-term oral steroids, chemotherapy, or an immune disorder)
* Requires immediate antiviral treatment or hospitalization as per the clinician's judgment
* Is allergic to trial medications
* Is scheduled for elective surgery or procedures requiring general anesthesia within the next two weeks
* Is co-infected with viruses of interest
* Received a live viral vaccine within the last 14 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 264 (Estimated)
Dates: Start 2026-01-02 (Estimated); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-04-24 (Estimated)

PRIMARY OUTCOMES:
time to recovery (defined as the first instance that a participant report feeling fully recovered) | Day 1 to Day 28
  The primary outcome is time to recovery (defined as the first instance that a participant report feeling fully recovered)

SECONDARY OUTCOMES:
All-cause emergency department (ED) visits | Day 1 to Day 28
  All-cause emergency department (ED) visits from randomization to 28 days, captured during participant daily diaries and corroborated with administrative data where possible, using administrative data holdings.
All-cause hospitalization visits | Day 1 to Day 28
  All-cause hospitalization visits from randomization to 28 days, captured during participant daily diaries and corroborated with administrative data where possible, using administrative data holdings.
All-cause death | Day 1 to Day 28
  All-cause death at 28 days from randomization to 28 days, captured during participant daily diaries and corroborated with administrative data where possible, using administrative data holdings.
Symptom severity obtained through daily diaries questionnaire | Day 1 to Day 28
  Symptom severity obtained through daily diaries questionnaire using the questions: "How is your general health? where 0 is poor and 5 is excellent and by rating symptoms, if present, as "No symptoms, mild, moderate, severe or very severe."
Quality of life obtained through the daily dairies using EQ-5D-5L | Day 1 to Day 28
  Quality of life obtained through the daily dairies using EQ-5D-5L
Costs and cost/QALY | Day 1 to Day 28
  Costs and cost/QALY assessed using data from participant daily diaries capturing health care use and treatment, combined with health-related quality of life measures.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Pinto, MD, Principal Investigator — Unity Health Toronto
Locations (1):
- Unity Health Toronto, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
Our team is dedicated to making data accessible to researchers upon request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: End of study (TBD) and upon request until 15years after study completion.
Access Criteria: Study PI
URL: https://upstreamlab.org/

REFERENCES:
- See also: study website — https://TreatResp.org
- See also: Lab website - Project page — https://upstreamlab.org/project/treatresp/